CLINICAL TRIAL: NCT07217600
Title: Efficacy and Safety of Ondansetron Orodispersible Film in Preventing Vomiting Induced by Moderately Emetogenic Risk Radiotherapy in Pediatric Patients With Malignant Tumors
Brief Title: Ondansetron Orodispersible Film for Vomiting Prevention in Pediatric Radiotherapy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yue Xie, Deputy Director, Chongqing University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CZLS2024304-A; ChiCTR2400093665 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2025-04-30; First posted 2025-10-16 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Radiotherapy-induced Nausea and Vomiting (RINV); Pediatric Cancer
MeSH Terms: conditions — Vomiting; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group QD (Experimental)
  Interventions: Drug: Ondansetron orodispersible film once
- group BID (Active Comparator)
  Interventions: Drug: Ondansetron orodispersible film twice

INTERVENTIONS:
Drug: Ondansetron orodispersible film once — Take ondansetron orodispersible film once 1-2 hours before each radiotherapy
  Arms: group QD
Drug: Ondansetron orodispersible film twice — Take ondansetron orodispersible film once before each radiotherapy , and once again 8 hours after the first dose.
  Arms: group BID

SUMMARY:
The goal of this study is to evaluate the antiemetic efficacy and drug safety of ondansetron orodispersible film in pediatric patients with malignant tumors who received moderate emetic risk radiation induced vomiting, and to formulate reasonable and effective clinical medication regimen for preventing vomiting caused by moderate emetic risk radiation in children with malignant tumor.

ELIGIBILITY:
Inclusion Criteria:

* Children with malignant tumors diagnosed by histopathology
* Age range: 1-14 years old (calculated from the day of signing the informed consent form)
* Weight >= 8Kg;
* Lansky functional status (LPS) score >= 50 (excluding posterior fossa syndrome)
* Be planned to undergo upper abdominal or craniospinal radiation therapy, and the upper abdominal irradiation should cover the anatomical area from the upper edge of the 11th thoracic vertebra to the lower edge of the third lumbar vertebra
* Radiotherapy is administered once daily, and the fractional dose is 1.8Gy, except for 1.5 Gy for whole abdominal radiotherapy
* The blood routine test must meet the following criteria: ANC >= 1.0 × 10^9/L (after discontinuation of G-CSF), PLT >= 50 × 10^9/L (without drug support or transfusion therapy), HGB >= 80g/L
* Biochemical tests must meet the following standards: total bilirubin <= 1.5 times ULN (upper limit of normal), ALT <= 2.5 times ULN, AST <= 2.5 times ULN, alkaline phosphatase ≤ 1.5 times ULN, serum albumin >= 2.5 g/dL, BUN and CRE <= 1.5 × ULN
* Expected survival period >= 3 months;
* The guardian of the child understands and signs the informed consent form, has good compliance, and cooperates with follow-up.

Exclusion Criteria:

* The nausea and vomiting caused by the surgery have not fully recovered if the subject has undergone a major surgery
* The patient has symptoms of central nervous system tumors such as cerebral edema and requires intervention with adrenal cortex hormones
* Participants who have participated in or are currently participating in other clinical studies within 4 weeks prior to the first use of the investigational drug (calculated based on the time of the last use of the investigational drug for those who have entered the follow-up period)
* Individuals allergic to 5-HT3 receptor antagonists or other excipients
* Joint use of apomorphine
* Congenital QT prolongation syndrome
* Severe gastrointestinal obstruction
* Other observers who affect the efficacy and adverse reactions
* Used other 5-HT3 receptor antagonists in the first 3 days of enrollment
* According to the researchers' assessment, there may be other factors that could force the subjects to terminate the study midway, such as suffering from other serious illnesses (including mental illnesses) that require concurrent treatment, severe abnormal laboratory test values, family or social factors that may affect the safety of the subjects or the collection of experimental data.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy in preventing vomiting between the two groups, as per the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 | From the first day of radiotherapy to 7 days after the end of radiotherapy
  Vomiting was divided into 5 grades according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0

SECONDARY OUTCOMES:
Adverse reaction rate | From the first day of radiotherapy to 7 days after the end of radiotherapy
The frequency of rescue treatments | From the first day of radiotherapy to 7 days after the end of radiotherapy
  Ratio of the number of rescue antiemetic uses to the number of radiotherapy fractions

CONTACTS AND LOCATIONS:
Overall Officials: Yue Xie, Principal Investigator — Chongqing University Cancer Hospital, Chongqing, China
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The initial data are available on request from the project leaders（344899525@qq.com），upon reasonable request.

REFERENCES:
- Available data/document: Study Protocol — https://www.chictr.org.cn/showproj.html?proj=253510